CLINICAL TRIAL: NCT07252128
Title: A Prospective Interventional Study Investigating the Effects of Brain Dynamic Audio Stimulation on Insomnia and Sleep Cycles in Healthcare Professionals
Brief Title: Effectiveness of Brain Dynamic Audio Stimulation for Improving Insomnia and Sleep Cycles in Healthcare Professionals
Acronym: BDAS-HP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chi Mei Medical Hospital (Other)
Responsible Party: Principal Investigator, Lin Hong-Min, Principal Investigator, Department of Family Medicine, Chimei Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11404-012; 11404-012 (Other: Chi Mei Medical Center)
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Sleep Disturbances and Insomnia
Keywords: Sleep Disturbance; Healthcare Workers; Non-Pharmacological Intervention; Brain Dynamic Audio Stimulation
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This is a single-group, pretest-posttest interventional study evaluating the effects of Brain Dynamic Audio Stimulation on sleep quality among healthcare professionals with subjective sleep disturbances. All participants receive the same intervention and serve as their own controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain Dynamic Audio Stimulation (Experimental): Participants in this experimental arm will receive Brain Dynamic Audio Stimulation (BDAS), a non-pharmacological auditory intervention designed to support sleep initiation and improve sleep quality. Each participant will use BDAS for 30 minutes once daily over two consecutive weeks in a controlled environment within Chi Mei Medical Center.
  The intervention will be delivered in a quiet and private setting to minimize external disturbances and ensure standardized conditions across sessions. The audio stimulation consists of frequency-modulated sound patterns intended to facilitate relaxation and support sleep onset.
  Pre- and post-intervention assessments will include the Insomnia Severity Index (ISI) as a subjective measure of sleep disturbance, as well as short-duration EEG-based sleep recordings. Objective sleep-related outcomes will be derived from EEG data, including sleep onset, sleep efficiency, and sleep stage distribution, in accordance with standardized sleep scoring criteria
  Interventions: Behavioral: Brain Dynamic Audio Stimulation

INTERVENTIONS:
Behavioral: Brain Dynamic Audio Stimulation — Participants will receive Brain Dynamic Audio Stimulation (BDAS), a non-pharmacological auditory intervention designed to support sleep initiation and improve sleep quality. The stimulation consists of frequency-modulated audio patterns delivered through headphones. Each participant will listen to a 30-minute session once daily for two consecutive weeks in a quiet, controlled environment.
  The intervention setting will be standardized to minimize external disturbances and ensure consistent delivery of the audio stimulation. The sound patterns are intended to facilitate relaxation and support the transition from wakefulness to sleep.
  Both subjective and objective sleep-related outcomes will be assessed before and after the intervention. Subjective sleep disturbance will be evaluated using the Insomnia Severity Index (ISI). Objective sleep parameters will be derived from short-duration EEG-based sleep recordings, including measures of sleep onset, sleep efficiency, and sleep stage distr
  Other Names: Brain Dynamic Audio

SUMMARY:
This study aims to evaluate the effectiveness of Brain Dynamic Audio Stimulation (BDAS) in improving sleep quality among healthcare professionals experiencing insomnia. Healthcare workers are frequently exposed to high occupational stress, irregular work schedules, and sleep disturbances, which may adversely affect mental well-being, cognitive performance, and clinical care.

Participants will use BDAS once daily for 30 minutes over a two-week period under standardized conditions. Both subjective and objective sleep-related outcomes will be assessed. Subjective sleep quality will be evaluated using the Insomnia Severity Index (ISI). Objective sleep parameters will be derived from short-duration EEG-based sleep recordings, including measures of sleep onset, sleep efficiency, and sleep stage distribution based on standardized scoring criteria.

This study seeks to determine whether audio-based neural entrainment through BDAS can facilitate sleep initiation and improve sleep efficiency in a real-world healthcare setting. As a non-pharmacological and non-invasive intervention, BDAS may offer healthcare professionals a safe and practical approach to managing insomnia and supporting overall well-being.

DETAILED DESCRIPTION:
Sleep disorders are recognized by the World Health Organization as a major global health issue, particularly among healthcare professionals exposed to high occupational stress and irregular work schedules. Although conventional pharmacological treatments for insomnia can be effective, they are often associated with adverse effects and the risk of dependence. Consequently, non-pharmacological approaches have gained increasing attention. Among these, audio-based brainwave entrainment has been proposed as a potential method to facilitate sleep initiation and stabilization through neural synchronization mechanisms.

This prospective interventional study adopts a single-group pretest-posttest design to evaluate the effects of Brain Dynamic Audio Stimulation (BDAS) on sleep quality in healthcare professionals. A total of 15 participants aged 20-65 years who report subjective sleep disturbances will be recruited from Chi Mei Medical Center, including nurses, physicians, therapists, and other allied healthcare workers. Exclusion criteria include recent use of hypnotics or psychotropic medications, diagnosed sleep disorders, and a history of major psychiatric, neurological, or severe chronic illnesses.

Participants will use BDAS once nightly for two consecutive weeks. Objective sleep-related data will be collected using short-duration EEG-based sleep recordings before and after the intervention to assess sleep onset, sleep efficiency, and sleep stage distribution, in accordance with standardized sleep scoring criteria. Subjective sleep outcomes will be evaluated using the Insomnia Severity Index (ISI). Pre- and post-intervention changes in ISI scores will be analyzed using paired statistical methods, while objective sleep parameters will be analyzed using appropriate comparative tests consistent with the exploratory nature of the study.

All study data will be de-identified and securely stored on password-protected institutional servers accessible only to authorized research personnel. Participation is voluntary, and participants may withdraw at any time without penalty. This study has been approved by the Institutional Review Board of Chi Mei Medical Center (IRB No. 11404-012; approval date: May 6, 2025).

ELIGIBILITY:
Inclusion Criteria:

* Licensed healthcare workers currently employed at Chi Mei Medical Center.
* Aged between 20 and 65 years.
* Experiencing subjective sleep disturbance or poor sleep quality for at least one month.
* Willing to participate in the Brain Dynamic Audio Stimulation sessions for two consecutive weeks.
* Able to provide informed consent and complete questionnaires and EEG assessments.

Exclusion Criteria:

* Current use of sedative-hypnotic medication, psychiatric medication, or other sleep-related pharmacotherapy.
* Diagnosed sleep disorders (e.g., obstructive sleep apnea, narcolepsy, restless legs syndrome).
* History of epilepsy, major psychiatric illness, or neurological disorder.
* Significant hearing impairment that interferes with audio stimulation.
* Pregnant or breastfeeding women.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) Score | From baseline (Day 0, prior to intervention) to post-intervention assessment (Day 14, after completion of two weeks of daily sessions).
  The Insomnia Severity Index (ISI) will be used to assess subjective insomnia severity before and after the intervention. The ISI is a validated 7-item self-reported questionnaire evaluating the severity, nature, and impact of insomnia symptoms, with each item rated on a 0-4 scale (total score range: 0-28). Higher scores indicate greater insomnia severity. The primary outcome is the within-participant change in total ISI score following Brain Dynamic Audio Stimulation, reflecting changes in perceived sleep disturbance among healthcare professionals.
Change in EEG-Derived Sleep Parameters | From baseline (Day 0, prior to intervention) to post-intervention assessment (Day 14, after completion of two weeks of daily sessions).
  Electroencephalography (EEG) will be used to derive objective sleep-related parameters before and after the Brain Dynamic Audio Stimulation intervention. Short-duration EEG-based sleep recordings will be analyzed to assess changes in sleep onset, sleep efficiency, and sleep stage distribution, based on standardized sleep scoring criteria. Pre- and post-intervention comparisons will be performed to evaluate objective changes in sleep patterns following the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Chi-Mei Medical Center, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the research team due to privacy protection of healthcare workers and institutional policy at Chi Mei Medical Center. Only aggregated and anonymized results will be published in academic journals or conferences.

REFERENCES:
- [Background] Abeln V, Kleinert J, Struder HK, Schneider S. Brainwave entrainment for better sleep and post-sleep state of young elite soccer players - a pilot study. Eur J Sport Sci. 2014;14(5):393-402. doi: 10.1080/17461391.2013.819384. Epub 2013 Jul 18. PMID 23862643
- See also: Chi Mei Medical Center Institutional Review Board — https://www.chimei.org.tw/main/cmh_department/59024/indexInternet.htm

DOCUMENTS (3):
  • Study Protocol (2026-01-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT07252128/Prot_003.pdf
  • Statistical Analysis Plan (2026-01-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT07252128/SAP_004.pdf
  • Informed Consent Form (2026-01-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT07252128/ICF_005.pdf